CLINICAL TRIAL: NCT06379035
Title: Blastocystis and Cryptosporidium Infection in Colorectal Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Hany Adly Ghaly, Dr Merna Hany Adly, Assiut University
Other Study IDs: Protozoa in CRC patients
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Blastocystis Infection; Cryptosporidium Infection; Colorectal Cancer
MeSH Terms: conditions — Blastocystis Infections; Cryptosporidiosis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ELISA / PCR — Multiplex PCR for confirmation of diagnosis of Blastocystis and Cryptosporidium infection.
  Enzyme linked immunosorbent assay (Elisa) for detection of :
  Different cytokines level in Colorectal cancer patients that may be involved in the tumor progression due to Blastocystis and Cryptosporidium infection.

SUMMARY:
1. Detect the prevelance of Blastocystis spp. and Cryptosporidium spp. among patients with colorectal cancer attending South Egypt Cancer Institute-Assiut University.
2. Detect the effect of Blastocystis and Cryptosporidium infection on various cytokines level in CRC patients that may be involved in the tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* The persons selected for the study are those who are:

  1. Colorectal cancer confirmed patients by imaging techniques (CT or MRI) and histopathological biopsy by Colonoscopy.
  2. Cooperative individuals attending South Egypt Cancer Institute - Assiut University of all ages and both sexes with confirmed diagnosis of CRC who agreed to be engaged in the study and were able to provide adequate samples.

CRC Patients will be divided into 4 groups:

Group 1: CRC patients without Blastocystis or Cryptosporidium infection. Group 2 : CRC patients with Blastocystis infection. Group 3 : CRC patients with Cryptosporidium infection. Group 4 : CRC patients with both Blastocystis and Cryptosporidium infection.

Exclusion Criteria:

* Patients having any type of tumors other than CRC. Patients taking anti-parasitic medications 2 weeks before sample collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Colorectal cancer confirmed patients by imaging techniques (CT or MRI) and histopathological biopsy by Colonoscopy.
  2. Cooperative individuals attending South Egypt Cancer Institute - Assiut University of all ages and both sexes with confirmed diagnosis of CRC who agreed to be engaged in the study and were able to provide adequate samples.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detect the prevelance of Blastocystis spp. and Cryptosporidium spp. among patients with colorectal cancer attending South Egypt Cancer Institute-Assiut University. | Baseline

SECONDARY OUTCOMES:
Detect the effect of Blastocystis and Cryptosporidium infection on various cytokines level in CRC patients that may be involved in the tumor progression. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Salma Mohammed Abd-ElRahman, Prof.Dr, Study Director — Assiut University; Rasha Abd-ElMonem Hassan, Prof.Dr, Study Director — Assiut University; Yasser Mohamed Mokhtar, Assis.Prof.Dr, Study Director — Assiut University

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Sulzyc-Bielicka V, Kolodziejczyk L, Jaczewska S, Bielicki D, Safranow K, Bielicki P, Kladny J, Rogowski W. Colorectal cancer and Cryptosporidium spp. infection. PLoS One. 2018 Apr 19;13(4):e0195834. doi: 10.1371/journal.pone.0195834. eCollection 2018. PMID 29672572
- [Background] Chan KH, Chandramathi S, Suresh K, Chua KH, Kuppusamy UR. Effects of symptomatic and asymptomatic isolates of Blastocystis hominis on colorectal cancer cell line, HCT116. Parasitol Res. 2012 Jun;110(6):2475-80. doi: 10.1007/s00436-011-2788-3. Epub 2012 Jan 26. PMID 22278727
- [Background] Ali SH, Ismail MAM, El-Badry AA, Abu-Sarea EY, Dewidar AM, Hamdy DA. An Association Between Blastocystis Subtypes and Colorectal Cancer Patients: A Significant Different Profile from Non-cancer Individuals. Acta Parasitol. 2022 Jun;67(2):752-763. doi: 10.1007/s11686-021-00508-y. Epub 2022 Jan 24. PMID 35067864
- [Background] Kumarasamy V, Kuppusamy UR, Samudi C, Kumar S. Blastocystis sp. subtype 3 triggers higher proliferation of human colorectal cancer cells, HCT116. Parasitol Res. 2013 Oct;112(10):3551-5. doi: 10.1007/s00436-013-3538-5. Epub 2013 Aug 10. PMID 23933809
- [Background] Sulzyc-Bielicka V, Kolodziejczyk L, Adamska M, Skotarczak B, Jaczewska S, Safranow K, Bielicki P, Kladny J, Bielicki D. Colorectal cancer and Blastocystis sp. infection. Parasit Vectors. 2021 Apr 14;14(1):200. doi: 10.1186/s13071-021-04681-x. PMID 33853659
- [Background] Abdou AG, Harba NM, Afifi AF, Elnaidany NF. Assessment of Cryptosporidium parvum infection in immunocompetent and immunocompromised mice and its role in triggering intestinal dysplasia. Int J Infect Dis. 2013 Aug;17(8):e593-600. doi: 10.1016/j.ijid.2012.11.023. Epub 2013 Jan 3. PMID 23291034
- [Background] Abd El-Latif NF, Kandil NS, Shamseya M, Elwany YN, Ibrahim HS. Role of Cryptosporidium spp in Development of Colorectal Cancer. Asian Pac J Cancer Prev. 2023 Feb 1;24(2):667-674. doi: 10.31557/APJCP.2023.24.2.667. PMID 36853318
- [Background] Kumarasamy V, Atroosh WM, Anbazhagan D, Abdalla MMI, Azzani M. Association of Blastocystis hominis with colorectal cancer: A systematic review of in vitro and in vivo evidences. World J Gastrointest Oncol. 2022 Mar 15;14(3):734-745. doi: 10.4251/wjgo.v14.i3.734. PMID 35321272
- [Background] Greige S, El Safadi D, Becu N, Gantois N, Pereira B, Chabe M, Benamrouz-Vanneste S, Certad G, El Hage R, Chemaly M, Hamze M, Viscogliosi E. Prevalence and subtype distribution of Blastocystis sp. isolates from poultry in Lebanon and evidence of zoonotic potential. Parasit Vectors. 2018 Jul 4;11(1):389. doi: 10.1186/s13071-018-2975-5. PMID 29973261